CLINICAL TRIAL: NCT05603585
Title: Attenuation of Sarcopenia Using Optimal Protein Supplementation and Early Exercise In Mechanically Ventilated Patients: A Pilot Randomized Controlled Trial (PIVOT)
Brief Title: Optimal Protein Supplementation and Early Exercise In Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/00201
Record Dates: First submitted 2022-09-19; First posted 2022-11-02 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-11

CONDITIONS: Nutritional Deficiency; Cachexia
MeSH Terms: conditions — Malnutrition; Cachexia

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to receive either standard feeding or optimised protein feeding based on random permuted blocks with age (≥65 years or < 65 years) and ICU site of recruitment as the stratification factors. The primary endpoint is difference in FSS between the two groups at Day 7.
Who Masked: Participant
Masking Description: The participants and their legally acceptable representative will not be made known of the experimental arms that the participant is allocated to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard care as per current ICU feeding regime.
- Interventional Group (Experimental): Optimal protein supplementation to achieve 80% protein adequacy through optimised protein supplementation. The protein supplementation will be increased/decreased based on the previous day's intake to achieve 80% adequacy each day by the dietician.
  Interventions: Dietary Supplement: Optimal protein supplementation to achieve 80% protein adequacy.

INTERVENTIONS:
Dietary Supplement: Optimal protein supplementation to achieve 80% protein adequacy. — Additional protein required and delivered by adding protein powder and given in bolus feeds
  Arms: Interventional Group

SUMMARY:
A Pilot Randomized Controlled Trial (RCT) will be conducted where where mechanically ventilated patients will be randomized to optimal protein (Achieve 80% protein supplementation adequacy with daily titration) versus standard protein feeding. Both groups will receive standard usual early exercise therapy.

Specific aim 1: To determine if optimal protein supplementation improves functional outcome of patients as measured by Functional Status Score (FSS) on Day 7.

Specific aim 2: To determine if optimal protein supplementation reduces muscle loss of patients at Day 7 as measured by the Rectus Femoris thickness and cross-sectional area (RFCSA) using skeletal muscle ultrasound.

Specific aim 3: To determine difference in functional recovery between groups using quality of life (QOL) scores and 6-minute walk distance at 3 months after hospital discharge.

The hypothesis is protein inadequacy can be overcome with optimized protein supplementation to reduce muscle loss/sarcopenia and functional impairment in ICU survivors.

DETAILED DESCRIPTION:
This study will be a prospective pilot randomized controlled trial. Collaboration will be between the National University Hospital (Medical, Surgical and Cardiothoracic ICUs), Centre for Healthy Aging, National University Health System (NUHS) and Physical Education & Sports Science, National Institute of Education (NIE). Patients admitted into these ICUs will be screened and those meeting the inclusion criteria will be approached for consent. If the patient is unable to consent, his/her legally acceptable representatives will be approached. This approach is routinely done in ICU studies. As with other ICU studies, potential difficulties in consenting and recruiting patients will be expected. To overcome this, all adult ICU patients at NUH will be included in the current study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and above.
2. Expected mechanical ventilation duration ≥ 48 hours.
3. Expected to stay in hospital for ≥ 4 days.

Exclusion Criteria:

1. Pregnant woman.
2. Amputation of either lower limbs.
3. Surgery of lower limb during the current admission.
4. 4. Any neurological/rheumatologic/orthopaedic/burn/trauma/physiological problem with feeding difficulties during 48h of intubation
5. Wheelchair-bound, walking aids and ADL-dependent.
6. Patient not able to feed by 48 hours AND not given parenteral feeding.
7. Patients on Continuous Renal Replacement Therapy.
8. Sepsis with poor prognosis.
9. Competing trial
10. Moribund within 48hours.
11. COVID-19 patients.
12. Declined to participate the study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional Status Score for ICU (FSS-ICU) | Day 1 of Randomisation; Day 7 of Randomisation; Day of ICU Discharge , approximately 14 days after ICU admission
  It is an ordinal score consisting of 5 activities (namely, Rolling in bed, Supine to Sit Transfer, Sit to Stand Transfer, Sitting Edge of Bed, Walking); each activity is scored from 0 to 7 to a total of 35. A higher score indicates a better functioning. It closely resembles Activities of Daily Living (ADL) and it is possible to even measure the pre-admission score. The FSS-ICU is measured at day 1 upon recruitment and compared to a one week period and to the time of discharge in intensive care to determine functional improvements at these time points.

SECONDARY OUTCOMES:
Rectus Femoris Cross-Sectional Area (RFCSA) and anterior thigh and rectus femoris thickness | Day 1 of Randomisation; Day 4 of Randomisation; Day 7 of Randomisation; Day of ICU Discharge , approximately 14 days after ICU admission
  RFCSA correlates well with quadriceps strength, measured by B-mode ultrasonography using linear transducer array. Pennation angle will also be calculated. The rectus femoris RFCSA and thigh thickness and pennation angle is measured at day 1 upon recruitment and compared to day 4 and then day 7 of study recruitment to determine changes in muscle loss.
Six-Minute Walk Test (6MWT) | 3 months post hospital discharge
  Feasible standard measure of exercise capacity
Clinical Frailty Index (CFI) | Day 1 of Randomisation; Day of ICU Discharge , approximately 14 days after ICU admission
  The CFI scoring is a scale from 1 to 9, 1 being very fit (best outcome) while 9 being terminally ill (worst outcome). The CFI is measured at day 1 upon recruitment and compared to point of ICU discharge to determine changes in frailty.
Blood Biomarkers | Day 1 of Randomisation; Day 4 of Randomisation
  The following cytokines; IL-6, IL-10, IL-12 and TNF-1α and MCP1, HMGB1 will be analysed via blood test to monitor inflammatory reactions
Indirect calorimetry (IC) | Day 1 to Day 7 of Randomisation (daily or till extubation)
  Gold standard for measurement of energy expenditure (EE)

CONTACTS AND LOCATIONS:
Overall Officials: Geetha Kayambu, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Participants ID will be coded as study participant ID. Only the PI and the study administrator will have access to the key between the code and participant ID.